CLINICAL TRIAL: NCT07056569
Title: Post-Marketing Clinical Follow-Up Trial to Evaluate the Performance and Safety of the Medical Device 047 TD Dermatitis Cream in Adults and Children With Atopic and Contact Dermatitis Symptoms Confirmed by Clinical Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biokosmes Srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 047 TD - BK2024
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Dermatitis, Contact; Dermatitis; Dermatitis, Chronic; Dermatitis, Eczematous; Dermatitis, Atopic Dermatitis
Keywords: Dermatitis; Atopic dermatitis; Contact dermatitis; Eczematous dermatitis
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis; Bronchiolitis Obliterans Syndrome; Eczema; Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 047_TD Dermatitis cream (Experimental): 047_TD Dermatitis cream formulation with a film-forming action intended for relieving dermatitis symptoms will be applied twice a day for 28 days on the affected skin zone.
  Interventions: Device: 047_TD Dermatitis cream twice a day for 28 days

INTERVENTIONS:
Device: 047_TD Dermatitis cream twice a day for 28 days — 047_TD Dermatitis cream will be applied twice a day for 28 days on the affected skin zone in sufficient amount of cream and let it dry.

SUMMARY:
The study aims to evaluate and confirm the performance of 047 TD Dermatitis cream in the improvement of eczematous dermatitis and contact dermatitis, throughout a reduction in disease severity and symptoms.

DETAILED DESCRIPTION:
The study hypothesis is to demonstrate that 047 TD Dermatitis cream creating a protective layer, on the area where it is applied, which defends the skin from external environmental factors.

The tool used in this research is a PMCF, a procedure which, through a scientific method of detection (one or more questionnaires to be submitted to a representative sample of patients related to the issue of the research), allows to collect, and subsequently analyze the data needed to study the relationships between different variables.

ELIGIBILITY:
Inclusion Criteria:

1. Male/ female > 6 months < 65 years
2. Patient diagnosed AD/CD
3. Patient with EASI max <16
4. Patient with IGA 1-3
5. Patient in good condition with no serious systemic disease

Exclusion Criteria:

1. Hypersensitivity to any 047_TD Dermatitis cream ingredients
2. Any other skin disease at the target area that would interfere the clinical assessment in the opinion of the investigator
3. Any other adjuvant therapy for AD/CD (UV therapy, probiotics, homeopathy etc.) within 30 days before Baseline as well as during the entire study
4. Any use of another topical emollient or other established treatment for AD/CD during the study at the site of flares (AD/CD lesions). Exception are usual hygienic products in the diaper area
5. A history of currently undergoing immunosuppressive drug therapy, chemotherapy, or radiation therapy
6. Drug abuser
7. Don't accept to attend the study procedures and processes as outlined in the protocol. Parents don't accept for the subject less 18th years old
8. Could not provide written informed consent or parents' informed consent to have their child participate in the study

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Performance measured by reduction of disease severity and symptoms | End of treatment - 28 days.
  The evaluation and confirmation of the performance of 047_TD Dermatitis cream in the improvement of eczematous dermatitis and contact dermatitis, through a reduction in disease severity and symptoms at 28 days of treatment, will be assessed by Investigator's Global Assessment (IGA) scores (successful threshold established as reduction of 1 point of the IGA score with respect to baseline value).

SECONDARY OUTCOMES:
Performance measured by reduction of disease severity and symptoms at 14 days | 14 days of treatment
  The evaluation and confirmation of the performance of 047_TD Dermatitis cream in the improvement of eczematous dermatitis and contact dermatitis, through a reduction in disease severity and symptoms at 14 days of treatment, will be assessed by Investigator's Global Assessment (IGA) scores (successful threshold established as reduction of 1 point of the IGA score with respect to baseline value).
Eczema improvement assessed by Eczema Area and Severity Index (EASI) score | Treatment day 14 and treatment day 28
  To evaluate the eczema improvement at 14 and 28 days of treatment with Eczema Area and Severity Index (EASI) score.
Pruritus improvement assessed by VAS | Treatment day 14 and treatment day 28
  Daily severity pruritus improvement measured by VAS improvement at 14 and 28 days of treatment.
Anti-itch effect measured by patient reported assessment | Day 1 of treatment
  Evaluated via subjective patient reported assessment the antiitch effect at day 1: immediate action (30sec-5min) and in 30 min.
Long lasting itch relief measured by patient reported assessment | Treatment day 14 and 28
  Evaluated via subjective patient/parent/caregiver reported assessment at day 14 and 28 - two times per day (8-10-12h)
Performance measured by improvement in the Quality of Life | Treatment day 1, 14 and 28
  Improvement in the quality of life of the subject related to their dermatitis will be assessed through the Dermatology Life Quality Index - Infant Dermatology Life Quality Index (DLQI/DLQC) questionnaire.
Subject adherence to treatment | From enrollment to the end of study on day 28
  Subject's adherence to treatment will be evaluated from daily diary compilation and product accountability.
Product usability | From enrollment to the end of study on day 28
  Assess through the subject's overall acceptability of the treatment.
Overall performance of the device | From enrollment to the end of study on day 28
  Assessment of the subject's and investigator's global evaluation of the performance of the product by measuring their satisfaction.
MD Safety evaluation | From enrollment to the end of study on day 28
  Evaluation of AE, SAE, ADE, SADE, ASADE, USADE incidence assessed by Investigator and reported according to the current legislation for the whole study period.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Studio Medico Pigatto Bersani, Milan
  - Poliambulatorio Verona, Verona
  - Studio Medico, Voghera

IPD SHARING:
Plan to Share IPD: No